CLINICAL TRIAL: NCT00637585
Title: A Comparison of Fexofenadine HCl 180 mg, Desloratadine 5 mg and Placebo in Suppression of Wheal and Flare Induced by Histamine
Brief Title: Fexofenadine HCl 180 mg, Desloratadine 5 mg and Placebo in Suppression of Wheal and Flare Induced by Histamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A_4145
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine

SUMMARY:
To examine the relative potency, onset of action and duration of action of fexofenadine HCl 180 mg (ALLEGRA) and desloratadine 5 mg (CLARINEX) as compared to placebo on skin wheals and flares induced by histamine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 12 to 55 years of age, may participate
* Positive histamine skin prick tests (or duplicate histamine skin prick test) with a summation flare (ΣF) greater than or equal to 20 mm larger than diluent control, and summation wheal (ΣW) greater than or equal to 6 mm larger than diluent control at the screening visit 1
* All female subjects must have a negative urine pregnancy test at the screening visit
* Female subjects who are sexually active will be expected to use one of the following birth control methods throughout the study (see Section 4.4)
* Subjects must be within 15% of normal body weight for height or a BMI less than 29.9 (based on NHLBI guidelines)
* Subjects willing and able to adhere to visit schedules and all study requirements
* All female subjects must have a negative urine pregnancy test at each treatment visit (Visit 2, 4, and 6).
* Continues to meet all inclusion and exclusion criteria

Exclusion Criteria:

* Asthma that requires treatment with medication other than an inhaled, short-acting beta agonist
* Signs and symptoms of currently active allergic disease (seasonal allergic rhinitis, perennial allergic rhinitis, episodic allergic rhinitis)
* Upper respiratory tract infection, sinusitis, asthma or flu-like symptoms within 2 weeks prior to visit 1
* Subjects who have dermatographism or other skin conditions which might interfere with the interpretation of the skin test results
* Subjects who are receiving immunotherapy
* Any excessive amounts of alcohol (no more than two drinks/day on average)
* Any excessive use of caffeine (more than six cups of coffee per day or equivalent)
* Any use of tobacco/nicotine products within 90 days of visit 1
* Any disease state or surgery known to affect the gastrointestinal absorption of drugs
* Known hypersensitivity to the investigational product or to drugs with similar chemical properties
* Subjects who will be visiting a tanning salon during the study
* Subjects who will need to use artificial tanning products during the study
* Night or variable shift workers during the study
* Pregnancy
* Breast-feeding
* History of hypersensitivity to the study medications or to drugs with similar chemical structures
* Treatment with other H1-receptor antagonists in the last year before study entry
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol (see Section 6.2)
* Treatment with any investigational product in the last 30 days before study entry
* No person or child of a person directly associated with the administration of the study may participate as a study subject
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Use of any of the following drugs within the time indicated prior to the first dosing visit:

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2002-12; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Size of change in summation skin flares from baseline will be measured. | Post-dose (20 min, 40 min, 60 min, and hourly through 12 hours with an additional 2 time points obtained at Hours 23 and 24)

SECONDARY OUTCOMES:
Size of change in summation skin wheals from baseline will be measured. | Post-dose (20 min, 40 min, 60 min, and hourly through 12 hours with an additional 2 time points obtained at Hours 23 and 24).

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States